CLINICAL TRIAL: NCT05439603
Title: A Phase 2 Study of ANC-501 in the Treatment of Adults With Major Depressive Disorder
Brief Title: ANC-501 in the Treatment of Adults With Major Depressive Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ancora Bio, Inc. d/b/a EmbarkNeuro, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ANC501D0005
Record Dates: First submitted 2022-06-21; First posted 2022-06-30 (Actual); Results first posted 2024-12-31 (Actual); Last update posted 2024-12-31 (Actual); Status verified 2023-02

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ANC-501 (Experimental): 50 mg/day
  Interventions: Drug: ANC-501

INTERVENTIONS:
Drug: ANC-501 — Five 10 mg capsules per day

SUMMARY:
A Phase 2 Study of ANC-501 in the treatment of adults with Major Depressive Disorder

DETAILED DESCRIPTION:
This is a single-arm, open-label Phase 2 study to assess the safety, tolerability, pharmacokinetics (PK), and activity of ANC-501 oral capsules as adjunctive treatment in subjects diagnosed with major depressive disorder (MDD)

ELIGIBILITY:
Inclusion Criteria:

* Adult male or female between 18 and 65 years of age, inclusive.
* Diagnosis of current episode of major depressive disorder (MDD) at least 8 weeks prior to screening, confirmed by Structured Clinical Interview for DSM-5 - Clinical Trials Version (SCID-5-CT).
* Have not responded to their current antidepressant therapy or to dose adjustment/treatment changes following a loss of response to their current antidepressant therapy.
* Receiving a stable dose of the same antidepressant (selective serotonin reuptake inhibitor [SSRI] or serotonin and norepinephrine reuptake inhibitor [SNRI], bupropion or trazodone monotherapy) for the current episode for at least 6 weeks of continuous treatment, which can include some or all of the screening period, with 4 weeks on a stable dose prior to day 1 and has an inadequate response (<50% improvement) using the MGH ATRQ.
* MADRS total score of ≥26 at screening and Day 1 (prior to dosing).
* 12-hour urine cortisol level >22.7 nmol/L(greater than or equal to 8.3 mcg/L).

Exclusion Criteria:

* Inadequate response to >2 prior ADTs (not including current antidepressant) of at least 6 weeks duration each for the episode current at screening.
* Medical history of bipolar disorder, schizophrenia, and/or schizoaffective disorder.
* Administration of drugs to treat psychiatric or neurologic conditions that have not been taken at a stable dose for at least 4 weeks prior to day 1.
* Significant findings on ophthalmic examination including, Best Corrected Visual Acuity (BCVA) worse than 20/30 or, in the opinion of the ophthalmologist or optometrist, any cataract that may become clinically significant and/or need surgical intervention during the course of the trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2022-09-19 (Actual); Primary Completion 2023-08-14 (Actual); Study Completion 2023-10-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Phil Perera, MD, Study Director — Ancora Bio, Inc. d/b/a EmbarkNeuro, Inc.
Locations (8):
- United States (8):
  - ATP Clinical Research, Orange, California
  - Florida Behavioral Medicine, Largo, Florida
  - Innovative Clinical Research, Inc., Lauderhill, Florida
  - Combined Research Orlando, Orlando, Florida
  - Clinilabs Drug Development Corporation, Eatontown, New Jersey
  - Clinilabs Drug development Corporation, New York, New York
  - Richmond Behavioral Associates, Staten Island, New York
  - Conrad Clinical Research, Edmond, Oklahoma

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This trial was conducted in 15 participants at 8 sites in the United States; 5 of the 8 trial sites enrolled subjects.
Pre-assignment Details: The total duration of participation is 20 weeks (up to 30 days screening, 8 weeks dosing, 8 weeks follow-up).
Groups:
- ANC-501: Participants were administered 50 mg ANC501 (5 x 10 mg) capsules orally once daily for 8 weeks in addition to their current stable dose antidepressant therapy (ADT).
Period: Overall Study
Arm/Group | ANC-501
Started | 15
Completed (One subject (out of the 13) completed all treatment visits and discontinued in the follow-up phase after last dose received.) | 13
Not Completed | 2
Not completed — met withdrawal criteria | 2

BASELINE CHARACTERISTICS:
Arm/Group | ANC-501
Number analyzed (Participants) | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.4 (13.25)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 11
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 10
  More than one race | 0
  Unknown or Not Reported | 1
Height [Mean (Standard Deviation); unit: cm] | 164.8 (7.87)
Baseline Weight [Mean (Standard Deviation); unit: kg] | 82.2 (15.64)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 30.2 (4.89)

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline (Day 1) to Day 56 in Montgomery-Asberg Depression Rating Scale (MADRS) Total Score.
Description: The MADRS was utilized as the primary efficacy assessment of the participant's level of depression. The MADRS consists of 10 items, all rated on a scale 0 to 6 with 0 being the "best" rating and 6 being the "worst" rating. The MADRS Total Score is the sum of ratings for all 10 items. Total MADRS score range is 0 to 60. A higher score indicates more severe depression.
Time Frame: Baseline (Day 1) to Day 56
Population: Efficacy population (N=13) consists of all subjects who received at least one dose of ANC501 and had completed treatment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ANC-501
Number analyzed (Participants) | 13
score on a scale | -17.5 (10.09)

2. Secondary Outcome: Mean Change From Baseline (Day 1) in Montgomery Asberg Depression Rating Scale (MADRS) Total Score at All Timepoints.
Description: The MADRS was utilized to assess the participant's level of depression. The MADRS consists of 10 items, all rated on a scale 0 to 6 with 0 being the "best" rating and 6 being the "worst" rating. The MADRS Total Score is the sum of ratings for all 10 items. Total MADRS score range is 0 to 60. A higher score indicates more severe depression.
Time Frame: Baseline (Day1), Day 8, Day 15, Day 29, Day 43, Day 56, and Day 70
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ANC-501
Number analyzed (Participants) | 13
score on a scale
  Day 8 | -11.9 (12.30)
  Day 15 | -15.6 (11.69)
  Day 29 | -18.6 (10.55)
  Day 43 | -17.8 (10.72)
  Day 56 | -17.5 (10.09)
  Day 70/FU | -18.8 (11.97)

3. Secondary Outcome: Percentage of Participants With Montgomery Asberg Depression Rating Scale (MADRS) Response.
Description: MADRS responder rate was defined as >=50% reduction in total score from Baseline (Day 1) to all time points. The MADRS consists of 10 questions, each rated on a 7-point scale, to stratify severity of depressive episodes. The MADRS total score is the sum of ratings for all 10 items. Total MADRS score range is 0 to 60. A higher score indicates more severe depression.
Time Frame: Baseline (Day1), Day 8, Day 15, Day 29, Day 43, Day 56, and Day 70
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | ANC-501
Number analyzed (Participants) | 13
Participants
  Day 8 | 6
  Day 15 | 6
  Day 29 | 8
  Day 43 | 9
  Day 56 | 7
  Day 70/FU | 7

4. Secondary Outcome: Percentage of Participants With Montgomery Asberg Depression Rating Scale (MADRS) Remission.
Description: MADRS remission rate was defined where total score was <=10 at all time points. The MADRS consists of 10 questions, each rated on a 7-point scale, to stratify severity of depressive episodes. The MADRS total score is the sum of ratings for all 10 items. Total MADRS score range is 0 to 60. A higher score indicates more severe depression.
Time Frame: Baseline (Day1), Day 8, Day 15, Day 29, Day 43, Day 56, and Day 70
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | ANC-501
Number analyzed (Participants) | 13
Participants
  Day 8 | 2
  Day 15 | 3
  Day 29 | 4
  Day 43 | 3
  Day 56 | 2
  Day 70/FU | 4

5. Secondary Outcome: Mean Change From Baseline (Day 1) to Day 56 in Hamilton Anxiety Scale (HAM-A) Total Score.
Description: The HAM-A was utilized as an assessment to rate participants level of anxiety. HAM-A is a 14-item questionnaire with each question rated on a 5-point scale with a total score of 0 to 56. The higher scores indicating more severe anxiety symptoms.
Time Frame: Baseline (Day 1) to Day 56
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ANC-501
Number analyzed (Participants) | 13
score on a scale | -7.6 (4.86)

6. Secondary Outcome: Mean Change in Clinical Global Impression-Severity (CGI-S) Score From Baseline (Day1) to Day 56.
Description: The CGI-S was utilized as an assessment for clinician to rate the severity of the patient's illness at the time of the assessment, relative to past experience with patients having the same diagnosis. CGI-S is a 7-point scale with response choices included: 0 = not assessed, 1 = normal, not at all ill, 2 = borderline mentally ill, 3 = mildly ill, 4 = moderately ill, 5 = markedly ill, 6 = severely ill, 7 = among the most extremely ill patients. The response at Day 56 was compared with the participants condition at Baseline prior to the first dose of study medication.
Time Frame: Baseline (Day1) to Day 56
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ANC-501
Number analyzed (Participants) | 13
score on a scale | -2.3 (1.25)

7. Secondary Outcome: Percentage of Participants With Clinical Global Impression-Improvement (CGI-I) Improvement
Description: The CGI-I was utilized as an assessment for clinician to rate the improvement of the patient's illness at the time of the assessment compared to patient's condition at admission of the trial. To perform this assessment, the study physician answered the following question: "Compared to his/her condition at admission to the project, how much has he/she changed?" This question is rated on a scale from 0 to 7, where a higher score indicates greater lack of improvement. Response choices included: 0 = not assessed, 1 = very much improved, 2 = much improved, 3 = minimally improved, 4 = no change, 5 = minimally worse, 6 = much worse, and 7 = very much worse. The response at a given visit was compared with the participants condition at Baseline prior to the first dose of study medication. A CGI-I improver was defined as a subject with a CGI-I score of "Very much approved" or "Much Approved".
Time Frame: Baseline (Day1), Day 8, Day 15, Day 29, Day 43, Day 56, and Day 70
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | ANC-501
Number analyzed (Participants) | 13
Participants
  Day 8 | 6
  Day 15 | 8
  Day 29 | 10
  Day 43 | 9
  Day 56 | 9
  Day 70 | 9

8. Secondary Outcome: Number of Participants With Clinical Global Impression-Improvement (CGI-I) Improvement
Description: The CGI-I was utilized as an assessment for clinician to rate the improvement of the patient's illness at the time of the assessment compared to patient's condition at admission of the trial. To perform this assessment, the study physician answered the following question: "Compared to his/her condition at admission to the project, how much has he/she changed?" This question is rated on a scale from 0 to 7, where a higher score indicates greater lack of improvement. Response choices included: 0 = not assessed, 1 = very much improved, 2 = much improved, 3 = minimally improved, 4 = no change, 5 = minimally worse, 6 = much worse, and 7 = very much worse. The response at a Day 56 was compared with the participants condition at Baseline prior to the first dose of study medication. A CGI-I improver was defined as a subject with a CGI-I score of "Very much approved" or "Much Approved".
Time Frame: Baseline (Day1) to Day 56
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | ANC-501
Number analyzed (Participants) | 13
Participants | 9

ADVERSE EVENTS:
Time Frame: Adverse events were reported from the signing of the informed consent until the last dose of ANC-501 with a safety follow-up of 8 weeks (+-3 days).
Description: One participant out of the 15 enrolled participants had one baseline AE that began prior to study drug dosing and continued during the study.
Arm/Group | ANC-501
All-Cause Mortality (participants affected / at risk) | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 11/15
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ANC-501 (N=15)
Tinnitus (Ear and labyrinth disorders) | 1 (1)
Elevated Amylase (Endocrine disorders) | 1 (1)
Elevated Lipase (Endocrine disorders) | 1 (1)
Bilateral Eye Disorder (Eye disorders) | 1 (1)
Blepharospasm (Eye disorders) | 1 (1)
Change in Cortical assessment per LOCS III >=0.5 in either eye compared to screening (Eye disorders) | 3 (3)
Change in Nuclear Opalescence per LOCS III >= 0.5 in either eye as compared to screening (Eye disorders) | 1 (1)
Right Eye Disorder (Eye disorders) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 3 (3)
Dry Mouth (Gastrointestinal disorders) | 2 (2)
Emesis (Gastrointestinal disorders) | 1 (1)
Flatulence (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (4)
Seasonal Allergies (Immune system disorders) | 1 (1)
Brown Vaginal Discharge (Infections and infestations) | 1 (1)
UTI (Infections and infestations) | 1 (1)
Back strain (Injury, poisoning and procedural complications) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Fracture Left Ankle (Injury, poisoning and procedural complications) | 1 (1)
Pain Left Ankle (Musculoskeletal and connective tissue disorders) | 1 (1)
Dizziness (Nervous system disorders) | 3 (3)
Burning While Urinating (Renal and urinary disorders) | 1 (1)
Increase Urinary Frequency (Renal and urinary disorders) | 1 (1)
Chest Congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Shortness of Breath (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sneeze (Respiratory, thoracic and mediastinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2023-03-07): https://cdn.clinicaltrials.gov/large-docs/03/NCT05439603/Prot_000.pdf
  • Statistical Analysis Plan (2023-09-29): https://cdn.clinicaltrials.gov/large-docs/03/NCT05439603/SAP_001.pdf